CLINICAL TRIAL: NCT01351545
Title: A Multicenter Access and Distribution Protocol for Unlicensed Cryopreserved Cord Blood Units (CBUs) for Transplantation in Pediatric and Adult Patients With Hematologic Malignancies and Other Indications
Brief Title: A Multicenter Access and Distribution Protocol for Unlicensed Cryopreserved Cord Blood Units (CBUs)
Status: Recruiting | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: 10-CBA; NCT01553461 (obsolete NCT alias)
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hematologic Malignancies; Inherited Disorders of Metabolism; Inherited Abnormalities of Platelets; Histiocytic Disorders; Acute Myelogenous Leukemia (AML or ANLL); Acute Lymphoblastic Leukemia (ALL); Other Acute Leukemia; Chronic Myelogenous Leukemia (CML); Myelodysplastic (MDS) / Myeloproliferative (MPN) Diseases; Other Leukemia; Hodgkin Lymphoma; Non-hodgkin Lymphoma; Multiple Myeloma/ Plasma Cell Disorder (PCD); Inherited Abnormalities of Erythrocyte Differentiation or Function; Disorders of the Immune System; Autoimmune Diseases; Severe Aplastic Anemia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Disease; Hodgkin Disease; Lymphoma, Non-Hodgkin; Autoimmune Diseases; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unlicensed CBU: The cohort includes recipients of any age receiving unlicensed cryopreserved cord blood units (CBUs) for designated indications.
  Interventions: Drug: A multicenter access and distribution protocol for unlicensed cryopreserved cord blood units (CBUs)

INTERVENTIONS:
Drug: A multicenter access and distribution protocol for unlicensed cryopreserved cord blood units (CBUs) — A multicenter access and distribution protocol for unlicensed cryopreserved cord blood units (CBUs) for transplantation in pediatric and adult patients with hematologic malignancies and other indications

SUMMARY:
This study is an access and distribution protocol for unlicensed cryopreserved cord blood units (CBUs) in pediatric and adult patients with hematologic malignancies and other indications.

DETAILED DESCRIPTION:
Principal Investigators:

The principal investigators (PIs) will be transplant physicians at all participating U.S. transplant centers.

Study Design:

This study is an access and distribution protocol for unlicensed cryopreserved cord blood units (CBUs) in pediatric and adult patients with hematologic malignancies and other indications.

Primary Objective:

The primary objective of this study is to examine the incidence of neutrophil recovery of ≥500/mm3 after cord blood transplantation in a multi-institution setting using CBUs that are not Food and Drug Administration (FDA) licensed.

Secondary Objectives:

In patients receiving a non-licensed CBU:

* Assess incidence of transmission of infection
* Assess incidence of serious infusion reaction
* Determine 1 year overall survival after cord blood transplantation
* Assess cumulative incidence of acute graft vs. host disease (GVHD) grades II to IV and grades III to IV
* Assess cumulative incidence of chronic GVHD
* Determine platelet engraftment of >20,000 mcL and >50,000 mcL

ELIGIBILITY:
Inclusion Criteria:

* Disorders affecting the hematopoietic system that are inherited, acquired, or result from myeloablative treatment
* Signed informed consent (and signed assent, if applicable) obtained prior to study enrollment
* Pediatric and adult patients of any age

Exclusion Criteria:

* Patients who are receiving only licensed CBUs
* Cord blood transplant recipients at international transplant centers
* Patients who are enrolled on another IND protocol to access the unlicensed CBU(s)
* Patients whose selected unlicensed CBU(s) will be more than minimally manipulated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recipients of unlicensed cryopreserved cord blood units who are being treated as U.S. transplant centers.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Estimated)
Dates: Start 2011-10; Primary Completion 2041-10 (Estimated); Study Completion 2041-10 (Estimated)

PRIMARY OUTCOMES:
Neutrophil recovery of ≥500/mm3 after cord blood transplantation | Cord blood engraftment occurs in weeks following transplant is defined as defined as ANC 500/mm3 and is analyzed at 60 days post-transplant.
  The primary objective of this access and distribution protocol is to examine the incidence of neutrophil recovery of ≥500/mm3 after cord blood transplantation in a multi-institution setting using CBUs that are not FDA licensed.
Neutrophil recovery of ≥500/mm3 after cord blood transplantation | Cord blood engraftment occurs in weeks following transplant is defined as defined as ANC 500/mm3 and is analyzed at 100 days post-transplant.
  The primary objective of this access and distribution protocol is to examine the incidence of neutrophil recovery of ≥500/mm3 after cord blood transplantation in a multi-institution setting using CBUs that are not FDA licensed.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Stefanski, MD, PhD, Study Chair — NMDP/CIBMTR
Locations (142):
- United States (142):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona (adults), Phoenix, Arizona
  - University of Arizona Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Children's Hospital of Los Angeles, Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - UCLA, Los Angeles, California
  - Children's Hospital and Research Center of Oakland, Oakland, California
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Sutter Medical Center, Sacramento, California
  - Rady Children's Hospital San Diego, San Diego, California
  - UCSF (adults), San Francisco, California
  - UCSF (Peds), San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Presbyterian St. Luke's/Colorado Blood Cancer Institute, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours - Alfred I. duPont Hospital for Children, Brandywine, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Medical Center, Gainesville, Florida
  - Nemours Children's Hospital - Mayo Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami (adult), Miami, Florida
  - University of Miami (peds), Miami, Florida
  - Niklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Florida Center for Pediatric Cellular Therapy, Orlando, Florida
  - Orlando Health Arnold Palmer Hospital for Children, Orlando, Florida
  - Orlando Health Cancer Institute Bone Marrow Transplant and Cellular Therapy, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University Health, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Indiana Blood & Marrow Transplantation, Beech Grove, Indiana
  - Indiana University/Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Westwood, Kansas
  - University of Louisville Hospital - James Brown Cancer Center, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Children's Hospital of New Orleans/LSUHSC, New Orleans, Louisiana
  - Greenebaum Cancer Center - University of Maryland, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Nih/Niaid, Bethesda, Maryland
  - NIH/NCI, Bethesda, Maryland
  - Nih/Nhlbi, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Univeristy of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - Washington University St. Louis, St Louis, Missouri
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson/Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Lake Sucess, New York
  - Cohen Children's Medical Center of New York, New Hyde, New York
  - New York University Langone Medical Center, New York, New York
  - New York Presbyterian Hospital at Cornell, New York, New York
  - Mount Sinai Medical Center - New York, New York, New York
  - Columbia University Medical Center - Morgan Stanley Children's Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Westchester Medical Center, New York, New York
  - Strong Memorial Hospital/University of Rochester, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Childrens Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Arthur G. James Cancer Hospital/The Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University/Doernbecher Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Cancer Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pennsylvania/Thomas Jefferson, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Transplant Institute, Sioux Falls, South Dakota
  - Methodist Healthcare Blood and Marrow Transplant Center, Memphis, Tennessee
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Sarah Cannon BMT Program, Nashville, Tennessee
  - VA Tennessee Valley Healthcare System, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Amarillo Blood and Marrow Transplant Program, Amarillo, Texas
  - Medical City Dallas, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Zachary & Elizabeth Fisher Bone Marrow Transplant Program (Brooke Army Medical Center), Fort Sam Houston, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital - Baylor Medical Center, Houston, Texas
  - Southwest Cancer Treatment & Research Center, Lubbock, Texas
  - The Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Healthcare System of San Antonio/Texas Transplant Institute, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - VA Puget Sound HCS, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin